CLINICAL TRIAL: NCT02100267
Title: A Study to Evaluate Efficacy and Safety of Methacholine Chloride Challenge Test in Diagnosis of Adult Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanwa Kagaku Kenkyusho Co., Ltd. (Industry)
Responsible Party: Sponsor
Purpose: Diagnostic
Other Study IDs: MC1001
Record Dates: First submitted 2014-03-24; First posted 2014-03-31 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Methacholine Chloride

ARMS (2):
- Asthma patients (Experimental)
  Interventions: Drug: Methacholine Chloride (SK-1211)
- Healthy volunteers (Experimental)
  Interventions: Drug: Methacholine Chloride (SK-1211)

INTERVENTIONS:
Drug: Methacholine Chloride (SK-1211) — Subjects received saline and 0.039-25 mg/mL of Methacholine chloride

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of Methacholine Chloride challenge test in diagnosis of adult asthma

ELIGIBILITY:
Inclusion Criteria:

* FEV1/forced vital capacity(FVC) must be 70% or more
* <10% decrease in FEV1 in response to inhalation of normal saline

Exclusion Criteria:

* Moderate airflow limitation (FEV1 < 60% predicted or < 1.5 L)
* Heart attack or stroke in last 3 months
* Uncontrolled hypertension, systolic BP>200, or diastolic BP>100

Ages: 20 Years to 64 Years | Sex: All
Age Groups: Adult
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of methacholine challenge test (Cutoff value of PC20: 8mg/mL) | Visit 2 (Day 1)
  Provocative concentration causing a 20% fall(PC20) will be captured once at visit 2.

CONTACTS AND LOCATIONS:
Locations (1):
- Showa University Clinical Research Center, Setagaya-ku, Tokyo, Japan